CLINICAL TRIAL: NCT06313632
Title: A Triple-Blind Randomized Controlled Trial of Erector Spinae Plane Block With Bupivacaine Versus Placebo in Patients Undergoing Medical Thoracoscopy
Brief Title: Erector Spinae Plane Block With Bupivacaine for Medical Thoracoscopy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: interim, lack of obvious benefit
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Udit Chaddha, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-23-01105
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pleural Disease; Postoperative Pain
Keywords: Thoracoscopy; Pleuroscopy; Regional Anesthesia; Erector Spinae Plane Block; Pain Control
MeSH Terms: conditions — Pleural Diseases; Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP with Bupivacaine Group (Experimental): Erector spinae plane block with bupivacaine.
  Interventions: Drug: Bupivacaine injection; Other: Monitored Anesthesia Care
- ESP with Placebo (Sham Comparator): Erector spinae plane injection with a placebo (normal saline).
  Interventions: Drug: Placebo; Other: Monitored Anesthesia Care

INTERVENTIONS:
Drug: Bupivacaine injection — Erector spinae plane block with bupivacaine (0.5%) 30 mL once
  Arms: ESP with Bupivacaine Group
Drug: Placebo — ESP with matching saline placebo
  Arms: ESP with Placebo
Other: Monitored Anesthesia Care — Standard monitored anesthesia care

SUMMARY:
PlAcebo versus erector spINae pLane block for mEdical ThoracoScopy Study (PAINLESS). This is a prospective triple-blind, randomized controlled trial that evaluates the efficacy of erector spinae plane block (ESPB) with Bupivacaine in reducing pain after medical thoracoscopy (MT) in addition to monitored anesthesia care vs monitored anesthesia care alone.

DETAILED DESCRIPTION:
This is a single-site prospect triple-blind, randomized controlled trial, that evaluates the efficacy of erector spinae plane (ESP) block with Bupivacaine in reducing pain after medical thoracoscopy (MT). The study aims to compare the effectiveness of ESP block with monitored anesthesia care (MAC) vs MAC alone for patients undergoing MT. Patient will be evaluated post operatively in the post anesthesia care unit and 24 hours after the procedure.

ELIGIBILITY:
Inclusion criteria:

* Referral for medical thoracoscopy
* Age ≥ 18

Exclusion criteria:

* Inability to provide informed consent.
* Study subject has any disease or condition that interferes with safe completion of the study including:

  * Allergic reaction to Bupivacaine.
  * Need for pleurodesis.
  * Allergies to lidocaine or other local anesthetics.
  * Pregnancy.
  * Advanced liver disease where the clinician deems the procedure unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 2 hours after the intervention
  Global chest pain score measured using the Visual Analog Scale (VAS) post-procedure in recovery. Participants will be asked to mark the level of their pain along a line, score ranges 0 (no-pain) to 100 (worst-imaginable pain), with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Change in the Numerical Rating Scale | At 2 hours post-intervention and 24 hours post-intervention
  Change in chest pain measured on the numerical rating scale post-procedure in recovery versus 24 hours post-procedure. This will be done using a numerical scale from 1 to 10 (1 = very mild pain, and 10 = very severe pain), with higher scores indicating greater levels pain. Data will be collected at the time of discharge from the recovery unit (2 hours post-intervention) vs 24 hours after.
Type of Analgesic use | within the first 24 hours after the intervention
  Type of Analgesic use within the first 24 hours after the intervention. The patient will be asked regarding the types of analgesics used (i.e. non-steroidal anti-inflammatories, opioids, etc.).
Number of Analgesic use | within the first 24 hours after the intervention
  Number of Analgesics used within the first 24 hours after the intervention. The patient will be asked regarding number of doses.
Dosage of Analgesic use | within the first 24 hours after the intervention
  Dosage of Analgesic used within the first 24 hours after the intervention. The patient will be asked regarding dose used.
Quality of Recovery-15 (QoR-15) Survey Score | within the first 24 hours after the intervention
  Compare quality of recovery 24 hours after the intervention. This will be evaluated with the QoR-15 questionnaire, scores range Minimum: 0 to Maximum: 150, with higher scores indicating a better outcome and better quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Udit Chaddha, MBBS, Principal Investigator — Principal Investigator
Locations (1):
- Mount Sinai West Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be processed by the research team. There is no plan to share IPD and only de-identified data will be collected.

REFERENCES:
- [Derived] Luebbert E, Salguero BD, Joy G, Salman S, Lo Cascio CM, Echevarria G, Chaddha U, Pai B H P. Benefits of Using Peripheral Nerve Blocks for Medical Thoracoscopy: A Retrospective Analysis. J Bronchology Interv Pulmonol. 2025 Mar 18;32(2):e1006. doi: 10.1097/LBR.0000000000001006. eCollection 2025 Apr 1. PMID 40099426